CLINICAL TRIAL: NCT03998891
Title: A Restricted Sodium Dietary Intake Reduces Hospital Admissions and Arrhythmic Burden in Patients Affected by Heart Failure With Reduced Ejection Fraction and Treated by Cardiac Resynchronization Therapy: Data From the SIRECART Registry
Brief Title: Sodium Intake in Failing Heart Patients.
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, principal investigator, University of Campania Luigi Vanvitelli
Other Study IDs: SecondUNI 20.06.2019
Record Dates: First submitted 2019-06-21; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Heart Failure; Salt; Edema
MeSH Terms: conditions — Heart Failure; Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- salt restricted diet: In this group the patients will received after CRTD a restricted (1500 grams/daily) salt intake.
  Interventions: Other: restricted dietary salt intake
- normal salt diet: In this group the patients will received after CRTD a normal (2500 grams/daily) salt intake.

INTERVENTIONS:
Other: restricted dietary salt intake — These patients after CRTd will receive a restricted dietary salt intake. To date, the salt intake will be 1500 grams daily.
  Groups: salt restricted diet

SUMMARY:
Patients with heart failure (HF) have an amelioration in clinical outcomes during a restricted dietary salt intake. To date, they experienced an amelioration of functional New York Association Heart (NYHA) class, reduction of hospital admissions, and mortality, in a percentage about 60%. However, these data have been not investigated in CRTd patients with HF under a condition of restricted vs. normal dietary salt intake. In the present study authors will evaluate clinical outcomes in patients treated by Cardiac Resynchronization Therapy with a defibrillator (CRT-d) and restricted dietary salt intake (group 1) in addition to conventional heart failure (HF) therapy vs. CRTd patients under conventional dietary salt intake and conventional HF therapy (group 2). The study will be conducted during a 12-months of follow-up, to evaluate the prognosis of CRTd patients treated with restricted (n 271) vs. a matched cohort of CRTd patients treated with normal salt dietary intake in addition to conventional HF therapy (n 288). Authors' opinion is that, restricted salt intake in addition to conventional HF therapy might significantly reduce body weight and heart chambers volumes in CRTd patients, leading to a significant improvement of ejection fraction and of the 6 minutes walking test (6MWT), and to a reduction of the arrhythmic burden. Consequently, restricted salt intake in addition to conventional HF therapy might reduce hospital admissions for heart failure worsening.

DETAILED DESCRIPTION:
Cardiac Resynchronization therapy with a defibrillator (CRTd) is a valid treatment for patients with heart failure and reduced left ventricle ejection fraction (HFrEF). Indeed, CRTd might induce an amelioration in New York Heart Association (NYHA) class, with a improvement of left ventricle ejection fraction (LVEF), and a reduction of hospital admissions for failing heart worsening. It is relevant to report that this ameliorative effect is seen only in a percentage about 70% of CRTd treated patients, that are called CRTd responders. However, about 30% of patients do not respond to CRTD, and they experience a worse clinical prognosis with an increasing trend toward heart failure (HF) disease progression, hospital admissions, and deaths. These patients are defined "CRTd non responders" . Actually, there is an increasing trend to find the mechanisms causing this therapeutic failure, such as a growing necessity to find new treatments to ameliorate CRTd effects, and to improve clinical outcomes in HFrEF patients with CRTd. In this setting, authors might speculate that salt and liquid retention represent a relevant pathogenic mechanism to cause worsening of NYHA class, with higher rate of hospital admissions for HF worsening and worse prognosis. Indeed, numerous studies reported the importance of a restricted vs. normal dietary salt intake in patients with HF to ameliorate clinical prognosis. Intriguingly, there are not studies investigating the effects of restricted dietary salt intake in failing heart patients with CRTd. Secondly, it is not well know how a restricted vs. normal dietary salt intake can affect clinical prognosis in CRTd patients. Therefore, the study hypothesis was that, a restricted dietary salt intake in addition to conventional anti-HF therapy as compared to the normal dietary salt intake in addition to conventional anti-HF drugs therapy might ameliorate heart function, and clinical outcomes in a population of HFrEF patients treated by CRT-d. Moreover, in this study authors will evaluate the effects of restricted vs. normal dietary salt intake in addition to conventional anti-HF in a population of failing heart patients treated by CRT-d. To date, in this study patients affected by HFrEF after CRT-d implant will be randomly divided in patients receiving restricted dietary salt intake plus conventional anti-HF therapy vs. patients under conventional dietary salt intake plus anti-HF therapy. In these patients authors will investigate at 12 months follow up all cause of deaths, cardiac deaths, hospitalizations for HF worsening, CRT-d responders rate, and the arrhythmic burden: atrial fibrillation (AF) events, ventricular tachycardia (VT) events, ventricular fibrillation (VF) events, internal cardioverter defibrillator (ICD) shocks, and strokes events.

ELIGIBILITY:
Inclusion Criteria:

* heart failure in NYHA 2-3 class;
* patients under optimal and full medical therapy for HF;
* patients treated with CRTd;
* patients without neoplastic diseases;
* patients without inflammatory sistemic diseases.

Exclusion Criteria:

* decompensated HF;
* unstable HF;
* patients without full anti-HF medical therapy;
* patients without indication to receive CRTd;
* patients with renal failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A population of patients affected by a stable and chronic heart failure in NYHA 2-3 class, and under optimal and full medical anti-HF therapy. These patients treated with CRTd will be aged between 18 and 75 years.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with heart failure worsening events | 12 months
  Authors will report by telephonic interviews, clinical visits and hospital discharge schedules the patients with HF worsening events.

CONTACTS AND LOCATIONS:
Locations (1):
- Raffaele Marfella, Naples, Italy